CLINICAL TRIAL: NCT04977635
Title: Biomarkers of Heterogeneity in Type 1 Diabetes: an Integrated Approach to Clinical and Metabolic Phenotyping of Individuals With Established Type 1 Diabetes
Brief Title: Biomarkers of Heterogeneity in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Diabeter Nederland BV (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL50314.042.15 / METc 2015/493; 3-SRA-2014-291-M-R (Other Grant/Funding Number: JDRF, Juvenile Diabetes Research Foundation)
Record Dates: First submitted 2021-07-13; First posted 2021-07-27 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes
Keywords: Heterogeneity; Biomarkers; C-peptide; Glucagon; Impaired awareness of hypoglycemia; Mixed meal tolerance test; Genetics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood samples will be collected in the following tubes: serum, Li-Hep, EDTA, EDTA P800, Paxgene RNA and Paxgene DNA.
  Fasting morning urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 600-cohort: Patients with long-term (> 5 years) type 1 diabetes aged 16 years and older
  As this is an observational study there is no intervention.

SUMMARY:
Biomarkers of heterogeneity in type 1 diabetes: establishment of a biobank and an integrated approach to clinical and metabolic phenotyping of individuals with established T1DM. In this project the investigators are searching for biomarkers in 600 patients with established (>5 years) diabetes. The inter-relation and patterns of expression in clinical, (auto)immune, metabolic, inflammatory and other parameters, and (potential) biomarkers are investogated. Blood and urine samples are collected annually (over 3 years) in standardized conditions and biobanked. In addition, 150 patients will undergo additional metabolic testing (such as mixed meal-tests).

DETAILED DESCRIPTION:
Identifying biomarkers of type 1 diabetes heterogeneity can help to stage the disease, and identify risks such as the early development of damage and complications.

Type 1 diabetes has long been considered to be an autoimmune disease in which failure of immune tolerance induces a specific immune attack on insulin-producing beta-cells. Recent research shows that the pathophysiology of type 1 diabetes is heterogeneous, involving various beta-cell-specific processes, different genetic predispositions, and several disease stages. It is very important to recognize this heterogeneity as it results in an accumulation of differences in outcomes during the course of the disease.

This heterogeneity requires further elucidation as a heterogeneous disease is likely to require multiple approaches to stop or cure the pathophysiological pathways. This underscores the need for more biomarkers to identify this heterogeneity, the different phases of disease and the effects of interventions and cures.

In many countries and research groups, data and samples from newly-diagnosed individuals (i.e. within the first 6 months after diagnosis) have been collected and studied. Fewer data and samples are available from patients with longer disease duration. This prompted JDRF to grant a strategic research agreement (SRA) to Diabeter and UMC Groningen. Both clinics have access to a substantial clinical database since 1998 with medical record data of > 3500 type 1 diabetes patients.

In this BIOMARKER project, the investigators intend to analyze hormonal, biochemical, immunological, inflammatory and psychological biomarkers of type 1 diabetes in patients with a disease duration of > 5 years. A sample repository (serum, plasma, urine, DNA, RNA) is established which is also accessible to other interested collaborators.

The collection currently includes:

* Fasting samples (serum, plasma, urine, DNA, RNA) from 600 patients with type 1 diabetes (> 5 years duration) taken annually at 3 timepoints
* Samples from 150 patients who underwent Mixed Meal Tolerance Tests (MMTT with 5 timepoints) at 2 occasions (1-year interval)
* Data from questionnaires on psychosocial burden, quality of life, neuropathy and hypoglycaemia completed by the patients
* Clinical datasets on their health, diabetes history, family history and clinical course during treatment

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes determined by either autoantibodies or based on clinical and historical data or both
2. At least 5 years (1825 days) of type 1 diabetes
3. Minimum age 16 years
4. Treated for type 1 diabetes at a diabetes center participating in this study
5. Subject understands study protocol and agrees to comply with it and has been able to read the patient information sheet, has had time to ask questions and get answers and gives signed informed consent.

Exclusion Criteria:

1. Non-type 1 diabetes
2. Patients with a duration of type 1 diabetes below 5 years
3. Patients under the age of 16 years
4. Pregnancy and breastfeeding, until 3 months (12 weeks) after childbirth or breastfeeding
5. On experimental medication or participating in other studies with conflicting goals and schedules
6. Diseases or conditions that the investigator/physician believes to be a contraindication to participate
7. Unwilling to be informed on incidental findings.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with >= 5 years duration of type 1 diabetes, age >= 16 years, treated for type 1 diabetes at a diabetes center participating in this study
Sampling Method: Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline remaining C-peptide production at 1 year and 2 years as measured by the Beckman ultrasensitive C-peptide assay | baseline, 1 year, 2 years
  Samples: fasting blood (serum)
Change in prevalence of impaired awareness of hypoglycaemia between baseline and 2-year timepoint as measured by adapted Clarke hypoglycaemia awareness survey | baseline, 2 years
  Correlation with C-peptide and clinical parameters
Genome-wide Association Study (GWAS) by Illumina 720k chip | cross-sectional: baseline
Assessment of glucagon response after stimulation with a mixed meal tolerance test as measured by the Mercodia glucagon assay (ELISA) | baseline
Change in patient-reported outcomes between baseline and 2 year timepoint as measured by WHO-5, PAID-20 and WHOQOL surveys | baseline, 2 years
  Quality of Life and problem areas in diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Henk-Jan Aanstoot, MD PhD, Principal Investigator — Diabeter Nederland BV; Bruce HR Wolffenbuttel, MD PhD, Principal Investigator — University Medical Center Groningen; Nel PH Geelhoed-Duijvestijn, MD PhD, Principal Investigator — Haaglanden Medical Center
Locations (3):
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Martine MC de Vries, Rotterdam
  - Haaglanden Medical Center, The Hague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Varkevisser RDM, Sas T, Aanstoot HJ; Dutch type 1 Biomarker group; Wolffenbuttel BHR, van der Klauw MM. Residual C-peptide is associated with new and persistent impaired awareness of hypoglycaemia in type 1 diabetes. J Diabetes Complications. 2024 Dec;38(12):108893. doi: 10.1016/j.jdiacomp.2024.108893. Epub 2024 Oct 22. PMID 39500130
- [Derived] Aanstoot HJ, Varkevisser RDM, Mul D, Dekker P, Birnie E, Boesten LSM, Brugts MP, van Dijk PR, Duijvestijn PHLM, Dutta S, Fransman C, Gonera RK, Hoogenberg K, Kooy A, Latres E, Loves S, Nefs G, Sas T, Vollenbrock CE, Vosjan-Noeverman MJ, de Vries-Velraeds MMC, Veeze HJ, Wolffenbuttel BHR, van der Klauw MM; Dutch Type 1 Diabetes Biomarker group. Cohort profile: the 'Biomarkers of heterogeneity in type 1 diabetes' study-a national prospective cohort study of clinical and metabolic phenotyping of individuals with long-standing type 1 diabetes in the Netherlands. BMJ Open. 2024 Jun 19;14(6):e082453. doi: 10.1136/bmjopen-2023-082453. PMID 38904129